CLINICAL TRIAL: NCT02760238
Title: Clinical and Molecular Epidemiology of Myeloproliferative Neoplasms (MPNs)
Brief Title: Myeloproliferative Neoplasms (MPNs) Patient Registry
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 15-9814 CE
Record Dates: First submitted 2016-03-24; First posted 2016-05-03 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Primary Myelofibrosis; Polycythemia Vera; Essential Thrombocythemia; Mastocytosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Juvenile; Chronic Eosinophilic Leukemia-not Otherwise Specified; Myelodysplastic-Myeloproliferative Diseases; Neoplasms; Leukemia, Myelomonocytic, Chronic
Keywords: myeloproliferative neoplasm; myelodysplastic syndrome; registry; leukemia; Bone Marrow Diseases; Hematologic Diseases; Neoplasms
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential; Mastocytosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Juvenile; Hypereosinophilic Syndrome; Myelodysplastic-Myeloproliferative Diseases; Neoplasms; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Myelodysplastic Syndromes; Leukemia; Bone Marrow Diseases; Hematologic Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of MPN: Patients with a myeloproliferative neoplasm (MPN) diagnosis:
  Atypical chronic myeloid leukemia (aCML), chronic eosinophilic leukemia-not otherwise specified (CEL NOS), chronic myelomonocytic leukemia (CMML), chronic neutrophilic leukemia (CNL), polycythemia vera (PV), essential thrombocythemia (ET), JMML, mastocytosis, MPN unclassifiable, myeloproliferative neoplasm/myelodysplastic syndrome unclassifiable (MPN/MDS unclassifiable), primary myelofibrosis (PMF), post-ET MF, post-PV MF, or (refractory anemia with ringed sideroblasts associated with marked thrombocytosis) RARS-T
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
The mandate of this MPN registry is to collect clinical information, including molecular results, from consenting patients with a variety of MPNs at different time points during the course of their disease.

DETAILED DESCRIPTION:
The myeloproliferative neoplasms (MPNs) are a group of rare hematological malignancies in which the bone marrow cells that produce the body's blood cells develop and function abnormally.

Despite the gains that have already been made in understanding and treatment of MPNs there is much that can still be learned. This registry will establish a clinical annotation database would help to better understand this group of diseases and to more effectively assign individual patients to the optimal therapy and so, improve their outcomes. This project will provide new insights on the molecular profiling of patients with MPN. It will be used as future resource for observational studies related to MPN.

The registry involves the collection of clinical information from patients with diagnosis of MPN at different time points during the course of their disease. The clinical data is collected following written informed consent from the Hematologic Malignancy tissue bank (UHN REB 01-0573C).

Data collected includes: a range of clinical measures, disease-associated factors, details of treatment and its results, complications during treatment, molecular and cytogenetic data, symptom assessment and survival outcome (up to 10 years).

Data will be collected prospectively and retrospectively, in both cases after obtaining written informed consent as per the study standard operating procedure (SOP).

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of one of the following myeloproliferative neoplasms (MPNs):

* Atypical CML (aCML)
* Chronic eosinophilic leukemia-not otherwise specified (CEL, NOS),
* Chronic myelomonocytic leukemia (CMML)
* Chronic neutrophilic leukemia (CNL),
* Essential thrombocythemia (ET),
* Juvenile myelomonocytic leukemia (JMML),
* Mastocytosis, MPN unclassifiable
* MPN/MDS unclassifiable,
* Primary myelofibrosis (PMF),
* Post-essential thrombocythemia myelofibrosis (post-ET MF),
* Post-polycythemia vera MF (post-PV MF)
* Refractory anemia with ringed sideroblasts associated with marked thrombocytosis (RARS-T)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at Princess Margaret Cancer Centre with an MPN diagnosis who consent to inclusion in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-04; Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Survival | Annually or at the time of transformation of disease, up to 10 years
  Survival of patients with MPN

SECONDARY OUTCOMES:
General patient characteristics will be captured from the Hematologic Malignancy tissue bank | Annually or at the time of transformation of disease, up to 10 years
  Type and phase of MPN, previous cancer history, age, sex
Disease risk score | Annually or at the time of transformation of disease, up to 10 years
  Risk stratification (IPSS, DIPSS and DIPSS)
  o Details of transformation to accelerated/phase phase disease
Quality of life - Neoplasm Symptom | Annually or at the time of transformation of disease, up to 10 years
  MPN-SAF TSS questionnaire
Co-morbidities | Annually or at the time of transformation of disease, up to 10 years
  HCT-CI
Physical symptoms of MPN | Annually or at the time of transformation of disease, up to 10 years
  Physical examination: Splenomegaly and hepatomegaly, ascites, EMS, ECOG
MPN treatment type received | Annually or at the time of transformation of disease, up to 10 years
  Medical therapies received
Transfusion dependence status | Annually or at the time of transformation of disease, up to 10 years
  Transfusion status
Current Blood Work | Annually or at the time of transformation of disease, up to 10 years
  CBC, INR, PT, APTT, fibrinogen, creatinine, ALP, ALT, AST, GGT, total bilirubin, LDH, urate, CRP, erythropoietin, hepatitis B and HIV
Identifying MPN driver mutations by using next generation sequencing. | Annually or at the time of transformation of disease, up to 10 years
  Next generation sequencing gene panel
Bone marrow transplant details (if received) | Annually or at the time of transformation of disease, up to 10 years
  Details of recipient (CMV status, ABO blood group)
  * Details of donor (gender, CMV status, ABO blood group)
  * Disease status at time of transplant (blood work disease status)
  * Transplant details (stem cell source, HLA matching, conditioning intensity & regimen, serotherapy, GVHD prophylaxis)
Bone marrow transplant complications (if received) | Annually or at the time of transformation of disease, up to 10 years
  Toxicities, engraftment and chimerism, GVHD, significant infections in the first 100 days
Portal hypertension | Annually or at the time of transformation of disease, up to 10 years
  Presence and details of ascites, GIT bleeding, esophageal & gastric varices, cirrhosis and portal hypertensive gastropathy
  o Endoscopy results
Pulmonary hypertension | Annually or at the time of transformation of disease, up to 10 years
  WHO classification, echocardiogram results, CNP, troponin, pulmonary function tests, 6 minute walk test distance, blood gas, treatment, complications
Thrombosis | Annually or at the time of transformation of disease, up to 10 years
  Details of thrombosis (type, site)
  o Treatment of thrombosis (type, duration)
Family history of MPN will be obtained from the patient record. | Annually or at the time of transformation of disease, up to 10 years
  Relative affected (e.g. daughter, uncle, mother), details of MPN (type, phase, treatment received)
Disease progression | Annually or at the time of transformation of disease, up to 10 years
  Risk stratification (IPSS, DIPSS and DIPSS)

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gupta, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be shared for REB approved research studies. Only the data necessary to achieve the study's aims will be shared and all data will be de-identified prior to sharing.
Time Frame: Continuing
Access Criteria: De-identified participant data may only be shared for REB approved research studies.

REFERENCES:
- [Derived] Medeiros JJF, Zeng AGX, Bansal S, Kim H, Chan-Seng-Yue M, Woo T, McLeod JL, Kothari S, Arruda A, Tsui H, Claudio JO, Maze D, Sibai H, Minden MD, Kennedy JA, Famulare CA, Rampal RK, Wang JCY, Dick JE, Gupta V. A Stem and Progenitor Cell-Derived Gene Expression Signature is Prognostic for Survival in Myelofibrosis. Blood. 2026 Jan 2:blood.2025030094. doi: 10.1182/blood.2025030094. Online ahead of print. PMID 41481381